CLINICAL TRIAL: NCT01127828
Title: Effects of Cultura Yoghurt on Symptoms Intestinal Flora and Immunological Changes in Patients With Irritable Bowel Syndrome(IBS)
Brief Title: Effects of Cultura Yoghurt in Irritable Bowel Syndrome (IBS) Patients on Intestinal and Immunological Changes
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Good Food Practice, Sweden (Industry)
Responsible Party: Magnus Simrén, Sahlgrenska University Hospital
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: U-05-008
Record Dates: First submitted 2010-05-20; First posted 2010-05-21 (Estimated); Last update posted 2010-05-24 (Estimated); Status verified 2010-05

CONDITIONS: Irritable Bowel Syndrome; Relief of Irritable Bowel Syndrome Symptoms; Quality of Life
Keywords: IBS (Irritable Bowel Syndrome); Probiotic yoghurt; Symptom severity
MeSH Terms: conditions — Irritable Bowel Syndrome

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Probiotic yoghurt (Cultura) (Active Comparator): Cultura yoghurt containing: L bulgaricus, S thermophilus
  Interventions: Other: Probiotic yoghurt (Cultura)
- Yoghurt with no probiotic (Placebo Comparator)
  Interventions: Other: Arla Yoghurt with no probiotic

INTERVENTIONS:
Other: Arla Yoghurt with no probiotic — two servings of 200 ml of investigational products per day
  Arms: Yoghurt with no probiotic
Other: Probiotic yoghurt (Cultura) — 200 ml per day
  Arms: Probiotic yoghurt (Cultura)

SUMMARY:
To determine the effect of cultura probiotic yoghurt on number of responders to treatment during 8 weeks of treatment in comparison to placebo. To determine the effect of cultura yoghurt on change in total score of (IBS) irritable bowel syndrome severity index during 8 weeks of treatment in comparison to placebo in IBS out patients.

DETAILED DESCRIPTION:
Recent research has shown taht probiotic may give positive effect on symptoms among patients with (IBS) Irritable Bowel Syndrome. The mechanism behind the positive effect are not known but a positive effect on different cytokines are a possible mechanism. Also effect on the large intestine bacterial mass could be of importance.

ELIGIBILITY:
Inclusion Criteria:

Signed consent to participate age 18-70 years IBS according to Rome II criteria

-

Exclusion Criteria:

1. Participation in a clinical study one month prior to screening visit and throughout the study.
2. Abnormal results of the screening laboratory tests clinically relevant for study participation, as judged by the investigator.
3. Other gastrointestinal disease(s) that explains the patient's symptoms, as judged by the investigator.
4. Other severe disease(s) such as malignancy, severe coronary disease, kidney disease or neurological disease, as judged by the investigator.
5. Symptoms indicating other severe disease(s) such as gastrointestinal bleeding, loss of weight or fever, as judged by the investigator.
6. Severe psychiatric disease as judged by the investigator.
7. Previous history of drug or alcohol abuse six months prior to screening.
8. Intolerance or allergy against milk products or gluten.
9. Use of other probiotic products (according to sponsor's list) 2 weeks prior to the study and throughout the study.
10. Consumption of antibiotic drugs 1 month prior to screening and throughout the study.
11. Consumption of cortisone, NSAID or other anti-inflammatory drugs on a regular basis 2 weeks prior to screening and throughout the study.
12. Pregnant or lactating or wish to become pregnant during the period of the study.
13. Lack of suitability for participation in the study for any reason as judged by the investigator.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2005-09; Primary Completion 2006-05 (Actual); Study Completion 2006-05 (Actual)

PRIMARY OUTCOMES:
Relief of IBS symptoms | 6 weeks intervention and 6 weeks follow up
  The primary endpoint of this study was the proportions of patients reporting adequate relief of their IBS symptoms at least 50 % of the weeks during the treatment period

SECONDARY OUTCOMES:
Effects on gastrointestinal and extraintestinal symptoms | September 2005 to May 2006
  effects of the investigational products on GI and extraintestinal symptoms assessed with the weekly IBS SSI questionnaire and the scores from the daily questions of the GI symptom questionnaire as weel as the effect on psychological symptoms and quality of life.

CONTACTS AND LOCATIONS:
Overall Officials: Magnus Simrén, Ass Prof, Principal Investigator — Medicine, Sahlgrenska University Hospital, S 413 45 Gothenburg, Sweden; Magnus Simren, Ass prof., Principal Investigator — Sahlgrenska hospital, Gothenburg, Sweden; Magnus Simrén, Ass proff, Principal Investigator — Medicine, Sahlgrenska University Hospital, S 413 45 Gothenburg, Sweden
Locations (1):
- Department of Internal Medicine, Sahlgrenska University Hospital, Gothenburg, Sweden